CLINICAL TRIAL: NCT02221362
Title: A Prospective, Noninterventional, Observational Study of Late-Onset Pompe Disease
Status: Terminated | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 701-901
Record Dates: First submitted 2014-08-06; First posted 2014-08-20 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2015-09

CONDITIONS: Late-onset Pompe Patients Untreated or Treated With rhGAA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples to be collected for exploratory research, Genetic/Genomic testing is optional requiring specific consent
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: No interventions

SUMMARY:
Study 701-901, a multicenter, multinational, longitudinal, non-interventional observational study in subjects, at least 18 years old, diagnosed with late-onset Pompe disease prospectively collects data to understand clinical progression in terms of respiratory function, symptomology, genotype, biochemistry, endurance and selected subject-reported measures for 24 weeks followed by a 240 week additional observation period for up to 100 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent after the nature of the study has been explained and prior to any study-related procedure
* Diagnosed with late-onset Pompe disease based on current or previous genomic testing and/or endogenous GAA activity
* At least 18 years of age at study entry
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Requires non-invasive ventilatory support while awake and in the upright position
* Concurrent disease, medical condition, or extenuating circumstance that, in the opinion of the investigator, might compromise study completion or data collection
* Unable to perform baseline efficacy assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Late-onset Pompe Disease patients untreated or treated with rhGAA
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the degree of change in respiratory and endurance endpoints over time in patients with Pompe disease | 264 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (24):
- Australia (3):
  - Westmead Hospital, Dept. of Genetic Medicine, Westmead, New South Wales
  - Women's and Children's Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
- Brazil (3):
  - Porto Alegre
  - Recife
  - Ribeirão Preto
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Greece (4):
  - Alexandroupoli
  - Athens
  - Larissa
  - Thessaloniki
- St. Vincent's University Hospital, Dublin, Ireland
- Poland (3):
  - Copernicus, St. Adalbert Hospital, Gdansk
  - Diamond Clinic, Krakow
  - Insitute of Psychiatry and Neurology, Warsaw
- Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei", Constanța, Romania
- Belgrade, Serbia
- National University Hospital, Singapore, Singapore
- Ljubljana, Slovenia
- Seoul National University Hospital, Seoul, South Korea
- Spain (3):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Mackay Memorial Hospital, Taipei, Taiwan